CLINICAL TRIAL: NCT07362004
Title: Validity and Reliability of an Immersive Virtual Reality Adaptation of the Timed Up and Go Test in Asymptomatic Young Adults
Brief Title: Virtual Reality-Based Timed Up and Go Test in Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_VR_TUG_ADAPTATION_1
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Functional Mobility; Virtual Reality-Based Functional Assessment
Keywords: Functional Mobility; Timed Up and Go Test; Virtual Reality; Immersive Virtual Reality; Validity; Reliability; Young Adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic Young Adults: Asymptomatic young adults aged 18-30 years undergoing conventional and immersive virtual reality-based Timed Up and Go assessments to evaluate feasibility, validity, and reliability.
  Interventions: Other: Clinical Assessments

INTERVENTIONS:
Other: Clinical Assessments — Participants will perform the Timed Up and Go test using an immersive virtual reality application developed for the Meta Quest 3 platform. The virtual environment digitally replicates the conventional test setup, including the starting position, turning point, and seating area. Test duration is automatically recorded by the system. The virtual reality-based assessment is designed to provide a standardized, objective, and reproducible evaluation of functional mobility and will be repeated to assess test-retest reliability.

SUMMARY:
Functional mobility encompasses the essential motor skills required for individuals to perform activities of daily living independently and safely. One of the most commonly used methods for assessing this parameter is the Timed Up and Go (TUG) test. The TUG test involves standing up from a chair, walking, turning, walking back three meters, and sitting down, and it is a measurement tool that has demonstrated high sensitivity and reliability in clinical practice for evaluating lower extremity function, mobility, and fall risk.

However, tests conducted in conventional clinical settings have limitations in terms of standardization due to examiner-related variability, environmental influences, and measurement subjectivity. These factors may lead to measurement errors, particularly when detecting small performance differences. Advances in virtual reality (VR) technology offer an innovative approach to the assessment and training of motor performance by recreating real-life scenarios in a three-dimensional and interactive manner. VR-based systems allow simultaneous observation of motor and cognitive processes while enhancing user motivation and engagement, thereby making the assessment process more dynamic. Recent studies have demonstrated that VR applications are effective tools in neurological rehabilitation, particularly in conditions such as multiple sclerosis (MS), for improving balance, walking speed, and functional mobility.

A review of the existing literature reveals that studies evaluating the validity and reliability of VR-based functional tests are limited. Moreover, to date, no study has specifically focused on the validity and reliability of the TUG test in an immersive VR environment for assessing lower extremity functional mobility. Therefore, this study aims to address a significant gap in the literature by being one of the first investigations to examine the validity and reliability of a VR-based version of the TUG test.

This study aims to determine the feasibility, validity, and reliability of the TUG test administered in an immersive VR environment in asymptomatic young adults aged 18-30 years. Additionally, the relationships between VR-based TUG outcomes and the 4-Meter Walk Test, the Four Square Step Test, and lower extremity muscle strength measurements will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years,
* Asymptomatic, with no musculoskeletal, neurological, or cardiovascular symptoms,
* Ability to perform activities of daily living independently,
* Visual, auditory, and vestibular functions suitable for virtual reality applications,
* Ability to understand and follow instructions in Turkish,
* Willingness to participate voluntarily in the study.

Exclusion Criteria:

* History of lower extremity injury, surgical intervention, or serious musculoskeletal condition within the past six months,
* Presence of vestibular disorders, balance impairment, visual or hearing impairments,
* Experiencing symptoms of "VR sickness," such as nausea, dizziness, or spatial disorientation during virtual reality applications,
* History of neurological, cardiovascular, or metabolic diseases,
* Regular participation in heavy exercise or professional sports activities,
* Cognitive impairment that prevents understanding of test instructions,
* Voluntary withdrawal from the study during the research process.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asymptomatic young adults aged 18-30 years who are able to perform activities of daily living independently and have no musculoskeletal, neurological, or cardiovascular conditions affecting functional mobility.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test - Virtual Reality (TUG-VR) | Baseline and 1-week follow-up
  This outcome measure will be used to assess functional mobility using an immersive virtual reality-based adaptation of the Timed Up and Go test. Test completion time will be automatically recorded by the system. Validity and reliability will be evaluated by comparison with the conventional Timed Up and Go test and repeated measurements performed one week apart.

SECONDARY OUTCOMES:
Timed Up and Go Test - Conventional | Baseline
  The conventional Timed Up and Go test will be administered to assess functional mobility and will be used as a reference measure for concurrent validity analysis.
4-Meter Walk Test | Baseline
  This test will be used to assess short-distance walking performance and gait speed. Results will be used for convergent validity analysis with the virtual reality-based Timed Up and Go test.
Four Square Step Test | Baseline
  This test will be administered to assess dynamic balance, agility, and directional change ability and will be used for convergent validity analysis.
Lower Extremity Muscle Strength | Baseline
  Lower extremity muscle strength will be measured using a handheld digital dynamometer to assess its relationship with functional mobility and virtual reality-based Timed Up and Go performance.
Participant Satisfaction | Baseline
  Participant satisfaction with conventional and virtual reality-based assessments will be evaluated using a 10-point numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Murat T İNANÇ, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maden C, Gozacan Karabulut D, Bagci B. Validity and reliability of an immersive virtual reality adaptation of the 6-minute pegboard and ring test. Hand Surg Rehabil. 2025 Feb;44(1):101981. doi: 10.1016/j.hansur.2024.101981. Epub 2024 Oct 30. PMID 39486588
- [Background] Massetti T, Trevizan IL, Arab C, Favero FM, Ribeiro-Papa DC, de Mello Monteiro CB. Virtual reality in multiple sclerosis - A systematic review. Mult Scler Relat Disord. 2016 Jul;8:107-12. doi: 10.1016/j.msard.2016.05.014. Epub 2016 May 21. PMID 27456884
- [Background] Maggio MG, Russo M, Cuzzola MF, Destro M, La Rosa G, Molonia F, Bramanti P, Lombardo G, De Luca R, Calabro RS. Virtual reality in multiple sclerosis rehabilitation: A review on cognitive and motor outcomes. J Clin Neurosci. 2019 Jul;65:106-111. doi: 10.1016/j.jocn.2019.03.017. Epub 2019 Mar 18. PMID 30898488
- [Background] Casuso-Holgado MJ, Martin-Valero R, Carazo AF, Medrano-Sanchez EM, Cortes-Vega MD, Montero-Bancalero FJ. Effectiveness of virtual reality training for balance and gait rehabilitation in people with multiple sclerosis: a systematic review and meta-analysis. Clin Rehabil. 2018 Sep;32(9):1220-1234. doi: 10.1177/0269215518768084. Epub 2018 Apr 13. PMID 29651873
- [Background] Kear BM, Guck TP, McGaha AL. Timed Up and Go (TUG) Test: Normative Reference Values for Ages 20 to 59 Years and Relationships With Physical and Mental Health Risk Factors. J Prim Care Community Health. 2017 Jan;8(1):9-13. doi: 10.1177/2150131916659282. Epub 2016 Jul 25. PMID 27450179
- [Background] Herman T, Giladi N, Hausdorff JM. Properties of the 'timed up and go' test: more than meets the eye. Gerontology. 2011;57(3):203-10. doi: 10.1159/000314963. Epub 2010 May 20. PMID 20484884